CLINICAL TRIAL: NCT02862509
Title: Effectiveness of Budesonide Nasal Instillation in a Vertex-to-floor Position in Chronic Rhinosinusitis Patients Underwent Endoscopic Frontal Sinus Surgery: a Randomized, Controlled Trial.
Brief Title: Effectiveness of Budesonide Nasal Instillation in a Vertex-to-floor Position
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Navarat Vatcharayothin, Principal Investigator, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE581299
Record Dates: First submitted 2016-07-16; First posted 2016-08-11 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Frontal Rhinosinusitis; Vertex to Floor Position
Keywords: Post-frontal sinus operation chronic rhinosinusitis patients; Budesonide nasal instillation; Vertex to floor position

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Budesonide nasal instillation (Experimental): budesonide(0.5mg/2ml) 1 respule plus normal saline solution 120ml instilled in vertex to floor position daily
  Interventions: Drug: Budesonide nasal instillation
- Normal saline nasal instillation (Placebo Comparator): Normal saline solution instilled in vertex to floor position daily
  Interventions: Drug: Normal saline nasal instillation

INTERVENTIONS:
Drug: Budesonide nasal instillation
  Arms: Budesonide nasal instillation
Drug: Normal saline nasal instillation
  Arms: Normal saline nasal instillation

SUMMARY:
o Chronic rhinosinusitis is one of the most common health issue affected American population. Surgery plays an important role in the patients who failed the medical treatment. The most difficult location to be operated endoscopically is the frontal sinus. Frontal sinus is also found to be one of the most common sinus for residual and recurrence after the operation. Intranasal steroid seems to be one of the most beneficent post-sinus surgery cares. The topical therapy can be delivered by many approaches. According to the standard clinical practice guideline and recommendations, intranasal corticosteroid spray is suggested. The technique proved to have greater distribution than standard intranasal spray is instillation of steroid nose drops. The head position for instillation of steroid nose drops proven to have a greater access to olfactory cleft and frontal area is Vertex-to-floor position.

ELIGIBILITY:
Inclusion Criteria:

* Chronic rhinosinusitis with frontal sinusitis patient
* Age ≥12
* Post-frontal sinus surgery with frontal sinus opening>3mm
* Satisfactory surgical technique: adequate sinus osteal drainage and mucosal sparing technique

Exclusion Criteria:

* Isolated frontal sinus surgery
* History of previous head and neck radiation
* Previous nasal or sinus operation
* Clinically significant deviated nasal septum
* History of paranasal sinus tumor
* Known immunocompromised Host
* History of budesonide allergy
* Cannot provide full flexion of the neck (cannot perform vertex-to-floor position)
* Post-randomization exclusion: Pathologic invasive fungal infection

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Total Sinonasal outcome test (SNOT) 20 score (validated Thai version) | three months

SECONDARY OUTCOMES:
Video-recorded nasal endoscope scoring: Modified Lund-Mackay Endoscopy Score(MLMES) | three months
Rhinological Sinonasal outcome test (SNOT) 20 score (validated Thai version) | three months

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok, Bangkok
  - Srinagarind Hospital, Khon Kaen, Changwat Khon Kaen

REFERENCES:
- [Result] Halawi AM, Smith SS, Chandra RK. Chronic rhinosinusitis: epidemiology and cost. Allergy Asthma Proc. 2013 Jul-Aug;34(4):328-334. doi: 10.2500/aap.2013.34.3675. PMID 23883597
- [Result] Blackwell DL, Lucas JW, Clarke TC. Summary health statistics for U.S. adults: national health interview survey, 2012. Vital Health Stat 10. 2014 Feb;(260):1-161. PMID 24819891
- [Result] Bhattacharyya N. Incremental health care utilization and expenditures for chronic rhinosinusitis in the United States. Ann Otol Rhinol Laryngol. 2011 Jul;120(7):423-7. doi: 10.1177/000348941112000701. PMID 21859049
- [Result] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. EPOS 2012: European position paper on rhinosinusitis and nasal polyps 2012. A summary for otorhinolaryngologists. Rhinology. 2012 Mar;50(1):1-12. doi: 10.4193/Rhino12.000. PMID 22469599
- [Result] Grobler A, Weitzel EK, Buele A, Jardeleza C, Cheong YC, Field J, Wormald PJ. Pre- and postoperative sinus penetration of nasal irrigation. Laryngoscope. 2008 Nov;118(11):2078-81. doi: 10.1097/MLG.0b013e31818208c1. PMID 18641522
- [Result] Musy PY, Kountakis SE. Anatomic findings in patients undergoing revision endoscopic sinus surgery. Am J Otolaryngol. 2004 Nov-Dec;25(6):418-22. doi: 10.1016/j.amjoto.2004.06.002. PMID 15547811
- [Result] Harvey RJ, Goddard JC, Wise SK, Schlosser RJ. Effects of endoscopic sinus surgery and delivery device on cadaver sinus irrigation. Otolaryngol Head Neck Surg. 2008 Jul;139(1):137-42. doi: 10.1016/j.otohns.2008.04.020. PMID 18585576
- [Result] Miller TR, Muntz HR, Gilbert ME, Orlandi RR. Comparison of topical medication delivery systems after sinus surgery. Laryngoscope. 2004 Feb;114(2):201-4. doi: 10.1097/00005537-200402000-00004. PMID 14755189
- [Result] Harvey RJ, Debnath N, Srubiski A, Bleier B, Schlosser RJ. Fluid residuals and drug exposure in nasal irrigation. Otolaryngol Head Neck Surg. 2009 Dec;141(6):757-61. doi: 10.1016/j.otohns.2009.09.006. PMID 19932850
- [Result] Hardy JG, Lee SW, Wilson CG. Intranasal drug delivery by spray and drops. J Pharm Pharmacol. 1985 May;37(5):294-7. doi: 10.1111/j.2042-7158.1985.tb05069.x. PMID 2862235
- [Result] Aoki FY, Crowley JC. Distribution and removal of human serum albumin-technetium 99m instilled intranasally. Br J Clin Pharmacol. 1976 Oct;3(5):869-78. doi: 10.1111/j.1365-2125.1976.tb00640.x. PMID 973982
- [Result] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Result] Snidvongs K, Dalgorf D, Kalish L, Sacks R, Pratt E, Harvey RJ. Modified Lund Mackay Postoperative Endoscopy Score for defining inflammatory burden in chronic rhinosinusitis. Rhinology. 2014 Mar;52(1):53-59. doi: 10.4193/Rhino13.056. PMID 24618629